CLINICAL TRIAL: NCT07103135
Title: Optimizing Accelerated TMS for Chronic Pain With Thompson Sampling
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: The Foundation for the Advancement of Clinical TMS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSYCH-2025-33814
Record Dates: First submitted 2025-04-24; First posted 2025-08-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a sham-controlled, single-blind, randomized study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study group (Experimental): Individuals with chronic pain
  Interventions: Device: MagVenture X100 Pro transcranial magnetic stimulation system

INTERVENTIONS:
Device: MagVenture X100 Pro transcranial magnetic stimulation system — The study intervention involves the use of the MagVenture X100 Pro transcranial magnetic stimulation system to deliver accelerated intermittent theta burst stimulation (aiTBS) to personalized targets within the somato-cognitive action network (SCAN) and action motor network (AMN) for the treatment of chronic pain.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of accelerated intermittent theta burst stimulation (aiTBS) targeting personalized nodes within the somato-cognitive action network (SCAN) and action motor network (AMN) for the treatment of chronic pain. The study will employ Thompson Sampling, a Bayesian reinforcement learning algorithm, to optimize stimulation site selection based on individual response patterns. This approach has the potential to revolutionize pain management by improving treatment accessibility through shortened timelines, addressing individual variations in pain networks through precision targeting, and potentially achieving more robust pain relief through accelerated neuroplasticity.

The specific aims of the study are:

1. To establish the relationship between SCAN and AMN connectivity and cognitive- affective pain symptoms.
2. To evaluate the efficacy of Thompson Sampling-optimized aiTBS across SCAN and AMN on affective and sensorimotor pain dimensions.
3. To identify fMRI connectivity biomarkers predictive of treatment response and remission.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years or older
* Ability to provide written informed consent
* Ability to read and to communicate verbally and in writing in English
* Chronic pain persisting for at least 12 months
* Pain refractory to oral pain medication (defined as failing at least two different medication classes)
* Average pain intensity of ≥5 on the Numerical Rating Scale (NRS) over the past two weeks
* Stable pain medication regimen for at least 4 weeks prior to enrollment
* Willing and able to attend all study visits and comply with study procedures

Exclusion Criteria:

* Current substance use disorder (except for nicotine or cannabis) as determined by DSM-5 criteria
* Active suicidal ideation with intent or plan as determined by the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Lifetime history of bipolar disorder, schizophrenia, or other psychotic disorder as determined by medical history
* Self-reported unstable medical conditions that would pose increased risks for TMS or MRI
* Pregnancy (as determined by urine pregnancy test) or planned pregnancy during the study period
* Contraindications to TMS, including:
* History of seizure or epilepsy
* Metallic implants in the head (excluding dental fillings)
* Cardiac pacemaker or other implanted medical devices
* History of significant head trauma
* History of intracranial surgery
* Medication that significantly lowers seizure threshold that cannot be safely held
* Contraindications to MRI, including:
* Claustrophobia
* Metallic implants or devices
* Inability to lie flat for the duration of the scan
* Current use of high-dose opioids (>90 morphine milligram equivalents daily)
* Participation in another clinical trial of an investigational medication or device within 30 days prior to enrollment
* Any condition that, in the investigator's opinion, would make it unsafe or difficult for the participant to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | 3 months
  measured by the Numerical Rating Scale (NRS) from baseline to after completion of the trial (approximately 3 months). For the NRS, the scores range from 0 to 10, where 0 indicates no pain (better outcome) and 10 is the worst pain that the participant can imagine (worse outcome)

SECONDARY OUTCOMES:
Change in pain intensity | Week 27
  NRS Scores
Change in sleep quality score | Week 21
  Measured by Garmin
Change in sleep time | Week 21
  Measured by Garmin
Adherence to the protocol and the tolerability of the study visits/procedures | Week 27
  Adherence to the protocol will be measured as participants completing at least 80% of the study activities. Tolerability: Measured by the average patient rating across study procedures. After completion of the study, we will collect feedback using a 5-point likert scale for measuring tolerability, we expect the average scores to be above 3.
Pain Catastrophizing Scale Score | Day 0
  The PCS is a 13-item questionnaire with each item scored 0-4, with higher scores indicating a worse outcome (higher tendency to catastrophize)
Pain Catastrophizing Scale Score | Week 15
  The PCS is a 13-item questionnaire with each item scored 0-4, with higher scores indicating a worse outcome (higher tendency to catastrophize)
Pain Catastrophizing Scale Score | Week 21
  The PCS is a 13-item questionnaire with each item scored 0-4, with higher scores indicating a worse outcome (higher tendency to catastrophize)
PROMIS Emotional Distress Score | Day 0
  15 items asking about anxiety and depression scored 1-5 with higher scores indicating worse outcomes (more severe symptoms of anxiety and depression)
PROMIS Emotional Distress Score | Week 15
  15 items asking about anxiety and depression scored 1-5 with higher scores indicating worse outcomes (more severe symptoms of anxiety and depression)
PROMIS Emotional Distress Score | Week 21
  15 items asking about anxiety and depression scored 1-5 with higher scores indicating worse outcomes (more severe symptoms of anxiety and depression)
Pain vigilance and awareness questionnaire (PVAQ) | Day 0
  The PVAQ is a 16-item questionnaire, where each item is scored as a six-point Likert scale that ranges from zero (never) to five (always), resulting in a sum score between zero and 80. Higher scores indicate worse outcomes (greater attention to pain)
Pain vigilance and awareness questionnaire (PVAQ) | Week 15
  The PVAQ is a 16-item questionnaire, where each item is scored as a six-point Likert scale that ranges from zero (never) to five (always), resulting in a sum score between zero and 80. Higher scores indicate worse outcomes (greater attention to pain)
Pain vigilance and awareness questionnaire (PVAQ) | Week 21
  The PVAQ is a 16-item questionnaire, where each item is scored as a six-point Likert scale that ranges from zero (never) to five (always), resulting in a sum score between zero and 80. Higher scores indicate worse outcomes (greater attention to pain)
Pain interference score on the Brief Pain Inventory (BPI) | Day 0
  The BPI is 11 items asking about pain sensations and interference with normal activity, all scored 0-10 with higher scores indicating worse outcomes (more pain or more interference due to pain)
Pain interference score on the Brief Pain Inventory (BPI) | Week 15
  The BPI is 11 items asking about pain sensations and interference with normal activity, all scored 0-10 with higher scores indicating worse outcomes (more pain or more interference due to pain)
Pain interference score on the Brief Pain Inventory (BPI) | Week 21
  The BPI is 11 items asking about pain sensations and interference with normal activity, all scored 0-10 with higher scores indicating worse outcomes (more pain or more interference due to pain)
Connectivity between SCAN and AMN connectivity on fMRI | Day 0
  The metric of connectivity will be the seeded correlation between the SCAN and the AMN
Changes in SCAN and AMN connectivity on fMRI | Week 21
  The metric of connectivity will be the seeded correlation between the SCAN and the AMN

CONTACTS AND LOCATIONS:
Overall Officials: Alexander B Herman, MD, PhD, Principal Investigator — University of Minnesota; David Darrow, Principal Investigator — University of Minnesota